CLINICAL TRIAL: NCT06719050
Title: Application and Evaluation of Telehealth-Based Chronic Disease Management for Type 2 Diabetes
Brief Title: Telehealth-Based Chronic Disease Management for Type 2 Diabetes
Acronym: T2DMTH
Status: Not yet recruiting | Type: Observational
Sponsor: Zeng Lin, Ph. D. (Other)
Responsible Party: Sponsor-Investigator, Zeng Lin, Ph. D., Deputy Director of Peking University Third Hospital Research Center of Clinical Epidemiology, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Other Study IDs: SF2024-2G-4097
Record Dates: First submitted 2024-11-28; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Type 2 DM

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (2):
- online + offline integrated management in the Internet hospital
- Routine offline management mode

SUMMARY:
This study will be conducted from enrollment until the end of the six-month follow-up period.

This study aims to assess the impact of the Internet hospital online + offline integrated chronic disease management model on patients with type 2 diabetes mellitus. It will also evaluate the economic impact of the model and identify the characteristics of the appropriate population for the model. Finally, it will develop a toolkit to help manage chronic diseases.

The study will include 1,636 patients with type 2 diabetes who did not reach the standard of control target of glucose, blood pressure or LDL at the endocrine outpatient clinic and inpatient wards of the Third Hospital of Peking University. We will collect information from participants before the study starts. And the patients will be followed up for 6 months from enrollment. The study management mode included online and offline integrated management in the Internet hospital, and routine offline management mode. After completing the enrollment and assessment, we will arrange outpatient follow-up and management according to the current status, doctor's requirements, and study subjects' needs.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old;
* Confirmed diagnosis of type 2 diabetes mellitus;
* Ability to use smartphones to participate in online diagnosis and treatment;
* Ability of the patient or relatives to assist the patient in self-monitoring of blood glucose;
* Failure to meet control targets: glycated hemoglobin ≥7. 0%, or LDL-C ≥ 2.6 mmol/L (and ASCVD or definite atherosclerosis with stenosis ≥ 1.8 mmol/L), or blood pressure > 130% and ≥ 1.8 mmol/kg. L), or blood pressure over 130/80 mmHg.

Exclusion Criteria:

* Mental illness, cognitive dysfunction;
* Other diseases and complex conditions (untreated tumors, heart disease within 3 months);
* Acute complications of diabetes, severe hyperglycemia, fasting glucose greater than 16.9 mmol / L, random glucose greater than 20 mmol / L. Diabetic ketoacidosis and hypoglycemic coma that are not suitable for online management of diabetes emergencies;
* Patients with severe chronic complications of diabetes in critical condition (blindness, vision deterioration, new onset of ASCVD symptoms);
* Those who are unsuitable for the study: infection, fracture, trauma, foot ulceration, edema, blindness, cardiovascular emergencies, coma, etc;
* Those who have not signed the informed consent form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients with type 2 diabetes who did not meet the control target of glucose, blood presure or LDL at the endocrine outpatient clinic and inpatient wards of the Third Hospital of Peking University.
Sampling Method: Probability Sample
Enrollment: 1636 (Estimated)
Dates: Start 2024-12-18 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients achieved all three targets (HbA1c < 7.0%, blood pressure < 130/80 mmHg and LDL-cholesterol < 2.6 mmol/L) | at 6±1 month from the enrollment

SECONDARY OUTCOMES:
patient adherence using 8-item Morisky Medication Adherence Scale (MMAS-8) | at 3±1 month from the enrollment
patient satisfaction using Visual Analogue Scale (VAS) | at 3±1 month from the enrollment
Hypoglycemic events | at 3±1 month from the enrollment
Acute complications | at 3±1 month from the enrollment
Hospitalization for any reason | at 3±1 month from the enrollment
blood glucose level | at 3±1 month from the enrollment
blood pressure assessment | at 3±1 month from the enrollment
Laboratory tests for blood lipid level (Low Density Lipoprotein-Cholesterol, LDL-C) | at 3±1 month from the enrollment
patient adherence using 8-item Morisky Medication Adherence Scale (MMAS-8) | at 6±1 month from the enrollment
patient satisfaction using Visual Analogue Scale (VAS) | at 6±1 month from the enrollment
blood glucose level | at 6±1 month from the enrollment
blood pressure assessment | at 6±1 month from the enrollment
diabetes self-management ability using Summary of Diabetes Self-Care Activities Questionnaire (C-SDSCA) | at 6±1 month from the enrollment
diabetes self-management ability using Confidence in Diabetes Management Self-Efficacy Scale (C-DMSES) | at 6±1 month from the enrollment
Direct Medical Cost | at 6±1 month from the enrollment
Laboratory tests for blood lipid level (Total Cholesterol, TC) | at 6±1 month from the enrollment
Laboratory tests for blood lipid level (Triglycerides, TG) | at 6±1 month from the enrollment
Laboratory tests for blood lipid level (Low Density Lipoprotein-Cholesterol, LDL-C) | at 6±1 month from the enrollment
Laboratory tests for blood lipid level (High Density Lipoprotein-Cholesterol, HDL-C) | at 6±1 month from the enrollment
Hypoglycemic events | at 6±1 month from the enrollment
Acute complications | at 6±1 month from the enrollment
Hospitalization for any reason | at 6±1 month from the enrollment

IPD SHARING:
Plan to Share IPD: Undecided